CLINICAL TRIAL: NCT02024217
Title: Phase II Study of Neoadjuvant Chemotherapy Wtih S1+Oxaliplatin (SOX) Regimen Followed by Chemoradiation Concurrent With S-1 in Patients With Potentially Resectable Gastric Carcinoma
Brief Title: Neoadjuvant Chemotherapy Plus Chemoradiation in Patients With Potentially Resectable Gastric Carcinoma
Acronym: NEWEAR
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhen Zhang, Chairman of Department of Radiation Oncology Fudan University Shanghai Cancer Center, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LAGCCS001
Record Dates: First submitted 2013-04-05; First posted 2013-12-31 (Estimated); Last update posted 2013-12-31 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — potassium oxonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chemoradiotherapy, S1, oxaliplatin (Experimental): chemoradiotherapy is given before surgical therapy,S1(Tegafur，Gimeracil and Oteracil Potassium Capsules) is given during radiation therapy and neoadjuvant chemotherapy, oxaliplatin is given during neoadjuvant chemotherapy.
  Interventions: Radiation: S1，oxaliplatin，radiation

INTERVENTIONS:
Radiation: S1，oxaliplatin，radiation — Radiation: 180 (cGy) /day, D1-5;S1: 50mg/m2,D1-5;
  Other Names: S1(Tegafur，Gimeracil and Oteracil Potassium Capsules)

SUMMARY:
To investigate the feasibility, safety and tolerability of Preoperative Chemoradiation in Patients With Localized Gastric Cancer. Primary endpoint: R0 resection rate. Secondary endpoint: resection rate, pathological complete regression (pCR), effectiveness and safety of regime, disease free survival(DFS) and overall survival(OS).

DETAILED DESCRIPTION:
The prognosis of gastric cancer is poor partially due to low R0 resection rate. Neoadjuvant chemoradiotherapy was reported to be effective in this setting by several phase II studies. The investigators aim to evaluate the efficacy and toxicity of neoadjuvant chemoradiotherapy in a prospective phase II study.

ELIGIBILITY:
Inclusion Criteria:

1.18 ≤ age ≤ 70, Male or Female; 2.Minimum life expectancy of 6 months; 3.Patients with localized, histologically confirmed gastric or gastroesophageal adenocarcinoma; 4.Patients must have a performance status of < 2 Eastern Cooperative Oncology Group (ECOG); 5.No prior major surgery of the stomach or radiation therapy to the stomach or immunotherapy or chemotherapy; 6.CT or MRI, endorectal ultrasonography (EUS), laparoscopic exploration are required to stage; 7.Without other benign diseases such as lung, kidney, liver infections; 8.Without participating other clinical trials; 9.Patient must sign an informed consent prior to study entry; 10.Patients must have adequate bone marrow function (defined as peripheral absolute granulocyte count of >1,500/µL, and platelet count of > 100,000/µL), adequate liver function (bilirubin <= 1.5 mg/dl), and adequate renal function (creatinine <= 1.5 mg/dl). 11)Patients without cardiac disease , severe uncontrolled diabetes, hypertension, cerebrovascular disease, or infection.

Exclusion Criteria:

1. Pregnant women are excluded from study entry due to the potential teratogenic effects of the study treatment;
2. Female patients who planed to have a baby;
3. Prior radiation therapy to the stomach, liver or kidney;
4. Dysfunction of important organs such as liver, kidney or heart; 5.Abnormalities of mental status;

6.Active coronary artery disease; 7.Cardiac arrhythmia, and need to receive medication therapy; 8.Severe uncontrolled hypertension; 9.Active clinical serious infection; 10.The known human immunodeficiency virus (HIV) infection history; 11.The known central nervous system diseases, including brain metastatic tumors; 12.Patients have had clinical clear gastrointestinal bleeding in 6 months; 13.Drug abuse; 14.Swallowing difficulties for drugs; 15.Poor compliance; 16.Presence of concurrent or previous malignancies (except for cervical carcinoma in situ or basal cell carcinoma of the skin); 17.Presence of peritoneal metastasis, distant organs or lymph nodes metastasis; 18.Presence history of major surgery in the past three months; 19.Poor tolerability; 20.Prior history of medication; 21.allergy for chemotherapeutic drugs.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-03; Primary Completion 2015-08 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
R0 resection rate | 6-8 Weeks
  6-8 weeks after Radiation therapy，we evaluate the lesion，if it is resectable，we will give surgical therapy，

SECONDARY OUTCOMES:
safety and tolerability of the treatment regimen | up to 10 weeks
  after neoadjuvant chemotherapy and chemoradiotherapy，we evaluate the side effects , and record the side effects

OTHER OUTCOMES:
resection rate | 6-8 Weeks
  6-8 weeks after Radiation therapy，we evaluate the lesion，if it is resectable，we will give surgical therapy，
disease-free survival | up to 36 months
  after surgical therapy，we followup the patients and stat the recurrence and death and calculate the disease-free survival
over-all survival | up to 36 months
  after surgical therapy，we followup the patients and stat the recurrence and death and calculate the over-all survival

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Result] Stahl M, Walz MK, Stuschke M, Lehmann N, Meyer HJ, Riera-Knorrenschild J, Langer P, Engenhart-Cabillic R, Bitzer M, Konigsrainer A, Budach W, Wilke H. Phase III comparison of preoperative chemotherapy compared with chemoradiotherapy in patients with locally advanced adenocarcinoma of the esophagogastric junction. J Clin Oncol. 2009 Feb 20;27(6):851-6. doi: 10.1200/JCO.2008.17.0506. Epub 2009 Jan 12. PMID 19139439
- [Derived] Liu X, Li G, Long Z, Yin J, Zhu X, Sheng W, Huang D, Zhu H, Zhang Z, Cai H, Huang H, Zhao G, Zhou Y, Zhang Z, Wang Y. Phase II trial of preoperative chemoradiation plus perioperative SOX chemotherapy in patients with locally advanced gastric cancer. J Surg Oncol. 2018 Mar;117(4):692-698. doi: 10.1002/jso.24917. Epub 2017 Nov 30. PMID 29194623